CLINICAL TRIAL: NCT03242200
Title: Assessing the Acceptability of the Use of a Mobile Health App Among Young Adult Female Survivors of Childhood Cancer: A Feasibility Study
Brief Title: Assessing the Acceptability of the Use of a Mobile Health App Among Young Adult Female Survivors of Childhood Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Villanova University (Other); Oncology Nursing Society (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: J1734; IRB00126543 (Other: JHM IRB)
Record Dates: First submitted 2017-07-17; First posted 2017-08-08 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2020-08

CONDITIONS: Childhood Cancer Survivor
Keywords: survivors of childhood cancer; young adult female; mobile app; questionnaire; health tracking

STUDY DESIGN:
Intervention Model Description: This project is a longitudinal one-group pilot study evaluating the use of a Mobile Health (mHealth) app intervention. This study will examine: 1) the amount/type of usage, 2 ) compliance with study evaluations and 3) the association of this mHealth app use with perceived self-efficacy in managing survivorship related needs, perceived health illness and health related quality of life. The study period will be nine months, with four measurement points to assess the study's outcomes: baseline, three, six, and nine months post initiation of the mHealth app.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mobile Health App (Other): Participants will be prompted to complete questionnaires.
  Interventions: Other: Mobile Health App

INTERVENTIONS:
Other: Mobile Health App — Mobile Health is a multi-featured app designed to enable participants to self-record and track their health and wellness. Participations will set up a profile and complete questionnaires. The app also records the amount of time and features of programs accessed.

SUMMARY:
The purpose of this research study is to understand if a mobile app is useful to assist young adult female survivors of childhood cancer in the self-management of survivorship-related needs.

DETAILED DESCRIPTION:
Survivorship related needs include managing lingering symptoms from treatment, how to keep a healthy lifestyle, social and medical issues, as well as other needs. The mobile health app that will be used in this study is the Health Storylines TM app developed by Self Care Catalysts Inc. The app can be used for an unlimited amount of time over nine months, which is how long the study will be conducted. The use of the Health Storylines TM app in this study is investigational.

Participation in this study starts with setting up a study specific profile on the app and entering information including email address, age, ethnicity/race, cancer diagnosis, as well as other optional information for the profile (example health goals or current health conditions). Participants will then be prompted by the app to complete three questionnaires about their ability to self-manage their survivorship-related needs, their perception of their survivorship-related illness symptoms and perceived health related quality of life. They will be prompted on the app to complete these questionnaires again at the 3, 6 and 9 month intervals of using the app. It will take about 20 minutes to complete the questionnaires at each measurement time. The only additional information that will be reported from the app for the study is the amount of time and features of programs accessed during the study period.

ELIGIBILITY:
Inclusion criteria are females who:

* Have been diagnosed with cancer before the age of 18 years
* Are between the ages 18 to 30 years
* Have been off treatment for at least six months
* Have a personal smart device to use for the app

Exclusion Criteria:

- None

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female survivors of childhood cancer
Enrollment: 30 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of mHealth app as measured by tracking all activities conducted on the app | Up to 2 years
  Assess the feasibility of the mHealth app as measured by tracking all activities of the patient-centered mHealth health tracking app, Health StorylinesTM, in young adult female survivors

SECONDARY OUTCOMES:
Adherence | Up to 2 years
  Assess the adherence to study procedures including baseline and follow-up assessments as measured by completion rates of required tasks
Self-Efficacy | Up to 2 years
  Determine the association between the amount of usage (in minutes), the frequency of usage number of times accessed) of the Health StorylinesTM mhealth app, and self-efficacy in young adult female survivors of childhood cancer.
Health Related Quality of Life | Up to 2 years
  Determine the association between the amount of usage (in minutes), the frequency of usage number of times accessed) of the Health StorylinesTM mhealth app and health related quality of life in young adult female survivors of childhood cancer
Perceived Illness | Up to 2 years
  Determine the association between the amount of usage (in minutes), the frequency of usage number of times accessed) of the Health StorylinesTM mhealth app and perceived illness in young adult female survivors of childhood cancer.

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Ruble, RN, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No